CLINICAL TRIAL: NCT06220214
Title: Contrast Enhanced Digital Mammography for Predicting Pathologic Complete Response After Neoadjuvant Chemotherapy
Brief Title: Neoadjuvant Therapy and Contrast-enhanced Mammography for Early Stage Breast Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Alison Stopeck (Other)
Responsible Party: Sponsor-Investigator, Alison Stopeck, Professor of Medicine, Stony Brook University
Organization: Stony Brook University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SBU-BC-NAC-CEDM; IRB2023-00508 (Other: Stony Brook IRB)
Record Dates: First submitted 2024-01-05; First posted 2024-01-23 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Locally Advanced Breast Cancer; Neoadjuvant Chemotherapy; HER2-positive Breast Cancer; Triple Negative Breast Cancer; TNBC, Triple Negative Breast Cancer
Keywords: cedm; cedbt; contrast-enhanced digital mammography; contrast-enhanced digital breast tomosynthesis; neoadjuvant chemotherapy
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- CEDM + CEDBT (Experimental): Participants undergo CEDM + CEDBT imaging after every 4-6 cycles of neoadjuvant chemotherapy prior to surgery (imaging may occur up to 2 times)
  Interventions: Diagnostic Test: CEDM; Diagnostic Test: CEDBT; Drug: Omnipaque 350mgI/mL Solution for Injection

INTERVENTIONS:
Diagnostic Test: CEDM — Contrast Enhanced Digital Mammography
Diagnostic Test: CEDBT — Contrast-Enhanced Digital Breast Tomosynthesis
Drug: Omnipaque 350mgI/mL Solution for Injection — Injection of an FDA approved iodinated contrast agent is required to undergo the imaging procedures. It is not the intent of the study to evaluate the contrast agent, but it will be administered at the time of experimental imaging.

SUMMARY:
The purpose of this study is to compare a special type of mammogram that uses a contrast agent called contrast-enhanced digital mammography with contrast-enhanced digital breast tomosynthesis (CEDM+CEDBT), with breast magnetic resonance imaging imaging (MRI) for predicting the effect of neoadjuvant chemotherapy on pathologic complete response rates. The device used to obtain CEDM+CEDBT images is called Siemens MAMMOMAT. This device produces two-dimensional (2D) images, as in a normal mammogram, but also collects additional images for digital breast tomosynthesis (DBT), which produces a three-dimensional (3D) image of the breast in the form of image slices. DBT allows the radiologist to "see through" the breast tissue for better detection and localization of breast cancer. By looking at both the CEDM images and the CEDBT images, a radiologist may be able to better detect residual breast cancer in a more cost-effective manner.

Participation may last up to 18 weeks.

Study procedures for this research are:

* Undergoing 1-2 mammograms during and/or after your chemotherapy, but before primary breast surgery.
* Before each mammogram, have a radiology technician inject a liquid contrast agent by inserting a needle into a vein. The chemotherapy port cannot be used to receive the contrast agent
* Let the research team record information from your medical record related to your condition and the treatment you receive.
* Give permission to collect leftover tissue from your diagnostic biopsy and breast surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis with either type of invasive locally advanced breast cancer regardless of hormone receptor or Her2 status
* Plan to receive at least 4 cycles of neoadjuvant chemotherapy ahead of definitive surgery

Exclusion Criteria:

* Pregnancy
* Allergy/sensitivity to contrast agent
* Decreased kidney function
* Diabetes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of (CEDM+CEDBT) to predict NAC treatment effects | Immediately after definitive breast surgery, up to 24 weeks
  The ability of CEDM + CEDBT to predict pathologic complete response to neoadjuvant chemotherapy, determined by histopathology evaluation of the resected breast

SECONDARY OUTCOMES:
Accuracy of (CEDM+CEDBT) to detect residual tumor compared with standard of care MRI | Immediately before definitive breast surgery
  Concordance between CEDM + CEDBT and standard of care MRI in quantifying residual tumor size

CONTACTS AND LOCATIONS:
Overall Officials: Alison Stopeck, MD, Principal Investigator — Stony Brook Cancer Center
Locations (1):
- Stony Brook Breast Center, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No